CLINICAL TRIAL: NCT00404170
Title: Assessing the Determinants of PD Progression - Long-term Dopamine Transporter Imaging in the PRECEPT Cohort
Brief Title: Assessing Imaging as a Tool in Monitoring and Predicting the Progression of Parkinson Disease
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Institute for Neurodegenerative Disorders (Other)
Collaborators: United States Department of Defense (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: Precept
Record Dates: First submitted 2006-11-22; First posted 2006-11-27 (Estimated); Last update posted 2022-07-05 (Actual); Status verified 2019-04

CONDITIONS: Parkinson Disease
Keywords: imaging; Parkinson; progression
MeSH Terms: conditions — Parkinson Disease; Disease Progression

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- B-CIT and SPECT imaging (Experimental): To assess B-CIT injection and SPECT scanning. Optional ongoing B-CIT SPECT imaging scans at follow-up visits
  Interventions: Drug: B-CIT and SPECT imaging

INTERVENTIONS:
Drug: B-CIT and SPECT imaging — Optional ongoing B-CIT SPECT imaging scans at follow-up visits

SUMMARY:
The purpose of this study is to investigate the utility of dopamine transporter imaging in monitoring and predicting the progression of Parkinson disease. This study will be performed in the PRECEPT cohort, an already existing cohort of 806 subjects recruited to participate in the study called, A Randomized, Double-Blind, Placebo-Controlled, Dose-Finding Study to Assess the Efficacy and Safety of CEP-1347 in Patients With Early Parkinson's Disease - (PRECEPT), sponsored by Cephalon and Lundbeck and coordinated by the Parkinson Study Group. The imaging data from this long-term PRECEPT follow-up study will allow us to evaluate the long-term progression of DAT loss in PD, the long-term follow-up of SWEDD subjects, the relationship between long-term clinical and imaging PD outcomes, and the relationship between long-term imaging outcomes and genetic and biochemical biomarkers of PD progression.

DETAILED DESCRIPTION:
The 800 early PD subjects in this study have already been evaluated clinically and have undergone longitudinal dopamine transporter (DAT) imaging with [123I] ß-CIT (baseline and 22 months). In Follow-up imaging will be performed at 24-month intervals (46 and 70 months following PRECEPT baseline). All scanning procedures will be performed at the Institute for Neurodegenerative Disorders (IND) using methods previously employed in the PRECEPT study.

Subjects willing to participate will travel to New Haven for their 46-month imaging visit. At IND a study coordinator and a neurologist will evaluate all subjects. The coordinator and neurologist will discuss the study procedures and evaluate the patient for eligibility. Written informed consent for the study will be obtained prior to performing any study-related procedures.

If eligible, participants will be injected with ß-CIT and 24 hours later an imaging procedure will be used to obtain pictures of brain activity using single photon emission computed tomography (SPECT). This 2-day procedure will be repeated at 70 months (following PRECEPT baseline).

ELIGIBILITY:
Inclusion Criteria:

* Subject was a participant in the PRECEPT clinical and imaging study
* Participant must be willing and able to comply with study procedures
* Participant must be willing and able to give informed consent.

Exclusion Criteria:

* The participant has a clinically significant clinical laboratory value and/or medical or psychiatric illness
* The participant has dementia (MMSE≤24)
* Pregnancy

Min Age: 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 396 (Actual)
Dates: Start 2006-11; Primary Completion 2014-07 (Actual); Study Completion 2014-07 (Actual)

PRIMARY OUTCOMES:
Assess progression of DAT loss during a 70 month interval | 70 months

CONTACTS AND LOCATIONS:
Overall Officials: Danna Jennings, MD, Principal Investigator — Institute for Neurodegenerative Disorders
Locations (1):
- Institute for Neurodegenerative Disorders, New Haven, Connecticut, United States

REFERENCES:
- See also: Institute for Neurodegenerative Disorders — http://www.indd.org